CLINICAL TRIAL: NCT00731458
Title: Prospective Comparison of Cirrus and Stratus Optical Coherence Tomography for Quantifying Retinal Thickness
Brief Title: Prospective Comparison of Cirrus Versus Stratus Ocular Coherence Tomography for Different Retinal Pathology.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Research to Prevent Blindness (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15606B
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Retinal Pathology
Keywords: OCT;; Cirrus;; Stratus;; macular thickness
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical coherance tomography ( Cirrus; Stratus) — Non-contact retinal thickness analyzer
  Other Names: OCT; Cirrus; Stratus

SUMMARY:
Ocular Coherence Tomography (OCT) is a non-invasive ophthalmologic test that uses reflected, unheated, non-concentrated visible light in order to scan and provide a 2-dimensional topographic analysis of the retina and optic nerve. It has wide diagnostic utility especially in patients with clinically significant macular edema, glaucoma, and other retinal eye diseases. At the University of Chicago, we have utilized the Stratus brand OCT (Carl Zeiss Inc) for the past 5 years. Recently we have acquired a beta version of the company's new model, the Cirrus HD-OCT (Carl Zeiss Inc.) which features improved resolution, shorter scanning time and a more user-friendly interface. The purpose of this study is to compare findings between the two models in patients with different common and uncommon eye diseases, including diabetic macular edema, glaucoma and age-related macular degeneration. We hypothesis that the Cirrus OCT is able to accurately quantify eye pathology compared to Stratus OCT.

ELIGIBILITY:
Inclusion Criteria:

* Any eye pathology that may cause macular edema.

Exclusion Criteria:

* Vitreous media opacities including dense cataracts, vitreous hemorrhage, and corneal opacities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seenu Hariprasad, M.D., Principal Investigator — University of Chicago

REFERENCES:
- [Background] Forooghian F, Cukras C, Meyerle CB, Chew EY, Wong WT. Evaluation of time domain and spectral domain optical coherence tomography in the measurement of diabetic macular edema. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4290-6. doi: 10.1167/iovs.08-2113. Epub 2008 May 30. PMID 18515567
- [Background] Gupta V, Gupta P, Singh R, Dogra MR, Gupta A. Spectral-domain Cirrus high-definition optical coherence tomography is better than time-domain Stratus optical coherence tomography for evaluation of macular pathologic features in uveitis. Am J Ophthalmol. 2008 Jun;145(6):1018-1022. doi: 10.1016/j.ajo.2008.01.021. Epub 2008 Mar 17. PMID 18343349